CLINICAL TRIAL: NCT00694655
Title: Human Immune Responses to Yellow Fever Vaccination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Sri Edupuganti, Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00009560; U19AI057266 (NIH)
Record Dates: First submitted 2008-05-19; First posted 2008-06-10 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Yellow Fever
Keywords: Yellow fever; Vaccine; Immunity; Yellow fever vaccine; CD8 T cell responses
MeSH Terms: conditions — Yellow Fever | interventions — Yellow Fever Vaccine; Leukapheresis; Biopsy, Fine-Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm A: Yellow Fever Vaccine in HLA-A202+ Participants (Experimental): HLA-A202+ participants receiving the Yellow Fever Vaccine plus post-vaccination blood draws.
  Interventions: Biological: Yellow Fever Vaccine
- Arm B: Yellow Fever Vaccine and Leukapheresis in HLA-A202+ Participants (Experimental): HLA-A202+ participants receiving the Yellow Fever Vaccine plus post-vaccination blood draws and leukapheresis.
  Interventions: Biological: Yellow Fever Vaccine; Procedure: Leukapheresis
- Arm C: Yellow Fever Vaccine and Fine Needle Aspirate in HLA-A202+ Participants (Experimental): HLA-A202+ participants receiving the Yellow Fever Vaccine plus post-vaccination blood draws and fine needle aspirate.
  Interventions: Biological: Yellow Fever Vaccine; Procedure: Fine-needle aspiration (FNA)
- Arm D: Yellow Fever Vaccine in HLA-A202- Participants (Experimental): HLA-A202- participants receiving the Yellow Fever Vaccine plus post-vaccination blood draws.
  Interventions: Biological: Yellow Fever Vaccine

INTERVENTIONS:
Biological: Yellow Fever Vaccine — Participants receive Yellow Fever Vaccine, at the FDA approved dose and route of administration.
  Other Names: YF-VAX; YFV-17D Yellow Fever Vaccine
Procedure: Leukapheresis — In leukapheresis blood is drawn and then the white blood cells are separated from the blood sample in a laboratory procedure. Once the white blood cells are returned the blood is returned back to the bloodstream of the participant who provided the sample.
  Arms: Arm B: Yellow Fever Vaccine and Leukapheresis in HLA-A202+ Participants
Procedure: Fine-needle aspiration (FNA) — In fine-needle aspiration a cell sample is collected using a needle and syringe. Fine-needle aspiration is typically used as a minimally invasive method of sample collection used to confirm a diagnosis.
  Arms: Arm C: Yellow Fever Vaccine and Fine Needle Aspirate in HLA-A202+ Participants

SUMMARY:
The goal of this study is to use the live attenuated Yellow Fever Vaccine (YFV) as a safe and effective model for viral infection to understand human immune response to viral antigens. Study participants will receive the yellow fever vaccine and participation in the study may be as short as one month or as long as one year, depending on immune responses.

DETAILED DESCRIPTION:
Yellow fever (YF) is a viral disease that is transmitted to humans through the bite of an infected mosquito. Yellow fever is a life-threatening infection that can result in hepatitis, renal failure and coagulation abnormalities, and in severe cases, death. Yellow fever was a major public health threat in the colonial United States in the 18th and 19th centuries.

Yellow fever is endemic in over 40 countries, and approximately 125 countries require proof of vaccination for entry by travelers at risk. An estimated 200,000 cases of yellow fever occur annually in South America and Africa, making it an important vaccine-preventable disease among travelers to endemic areas. Yellow fever can be prevented by vaccination with the Yellow Fever Vaccine. Currently, the Centers for Disease Control and Prevention (CDC) and the World Health Organization (WHO) recommend yellow fever vaccination for persons ≥ 9 months of age who are traveling to or living in a yellow fever endemic area.

The Yellow Fever Vaccine is considered to be one of the safest and most effective viral vaccines ever developed. Yellow Fever Vaccine is known to stimulate broad-spectrum immune responses, including cytotoxic T cells, and Th1 and Th2 responses, as well as neutralizing antibody titers that can persist for up to 30 years, after a single vaccination. Despite the great success of this empiric vaccine, there has been relatively little understanding of the mechanisms by which Yellow Fever Vaccine induces such robust protective immune responses. The researchers hope to apply the best contemporary methods in immunology, genomics, and proteomics to characterize in detail a successful immune response to Yellow Fever vaccination. This characterization should identify new immunologic predictors that could serve as surrogates for future vaccine efficacy studies. In addition, these findings could guide development of a safer yellow fever vaccine (or the derivation of safer alternative vaccination regimens using the currently available vaccine).

This study plans to recruit both travelers to yellow fever endemic areas as well as non-travelers for participation. Healthy participants will be enrolled into four study arms. Arm enrollment is determined by Human Leukocyte Antigen (HLA) type, current needs of the lab and/or willingness to participate in sampling procedures. All participants receive Yellow Fever Vaccine on Day 0 at the FDA-approved dose and route of administration. Post-vaccination procedures are determined by arm assignment. Participants will be followed for up to 360 days post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and give informed consent
2. Age 18-45 years
3. Participant agrees not to take any live vaccines 30 days before or after (14 days for inactivated, including coronavirus disease 2019 (COVID-19) vaccination) yellow fever vaccination
4. Women of child bearing potential must agree to use effective birth control throughout the duration of the study. A negative urine pregnancy test must be documented prior to vaccination. Participants who have a history of surgical sterilization or post-menopausal status >1 year, are not required to have a pregnancy test.

Exclusion Criteria:

1. Prior receipt of a yellow fever vaccine
2. Lived in a country/area which is endemic for yellow fever
3. Travel to country/area which is endemic for yellow fever. Subject to investigator discretion
4. History of previous yellow fever, West Nile, Dengue, St. Louis encephalitis, Japanese encephalitis vaccination or infection
5. Any history of allergy to eggs, chicken or gelatin or to any previous vaccine
6. A history of a medical condition resulting in impaired immunity (such as HIV infection, cancer, particularly leukemia, lymphoma, use of immunosuppressive or antineoplastic drugs or X-ray treatment). Persons with previous skin cancers or cured non-lymphatic tumors are not excluded from the study
7. History of HIV infection
8. Active Hepatitis B or Hepatitis C infection
9. COVID-19 infection in the last 30 days. Symptoms of COVID-19 must be completely resolved before yellow fever vaccine receipt.
10. History of any chronic medical conditions that are considered progressive (ex, diabetes, heart disease, lung disease, liver disease, kidney disease, gastrointestinal diseases and uncontrolled hypertension). Use of systemic immunosuppressive medications (ex, prednisone) for 2 weeks or more in the past 3 months
11. History of excessive alcohol consumption, drug abuse, psychiatric conditions, social conditions or occupational conditions that in the opinion of the investigator would preclude compliance with the trial
12. Thymus gland problems (such as myasthenia gravis, DiGeorge syndrome, thymoma) or removal of thymus gland or history of autoimmune disorder
13. Recipient of a blood products or immune globulin product within 42 days of the vaccination visit. Participants who received COVID monoclonal antibodies (mAbs) for treatment are not excluded
14. Pregnant women and nursing mothers or women who are planning to become pregnant for the duration of the study
15. Any condition in the opinion of the investigator that would interfere with the proper conduct of the trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 239 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Magnitude of Yellow Fever Virus (YFV) specific T Cell Responses | Day 0 (day of vaccination), Day 7, Day 14, Day 21, Day 28, Day 90, Day 180, Day 360
  The characterization of Yellow Fever Vaccine specific adaptive immune response will be examined as the magnitude of YFV-specific T cell responses. The schedule of follow up visits depends on if participants test positive for human leukocyte antigen (HLA) A202 and the different immune system responses that the study team is examining at the time when each participant enrolls.
Quality of YFV-specific T Cell Responses | Day 14, Day 21, Day 28, Day 90, Day 180, Day 360
  The characterization of Yellow Fever Vaccine specific adaptive immune response will be examined as the quality of YFV-specific T cell responses. The schedule of follow up visits depends on if participants test positive for HLA-A202 and the different immune system responses that the study team is examining at the time when each participant enrolls.

SECONDARY OUTCOMES:
Characterization of Cytomegalovirus (CMV) | Day 0 (day of vaccination), Day 21, Day 180
  Characterization of CMV CD8 T cells will be performed. The schedule of follow up visits depends on if participants test positive for HLA-A202 and the different immune system responses that the study team is examining at the time when each participant enrolls.
Phenotypic Analysis of Cytomegalovirus (CMV) | Day 0 (day of vaccination), Day 21, Day 180
  Phenotypic analysis of CMV CD8 T cells will be performed. The schedule of follow up visits depends on if participants test positive for HLA-A202 and the different immune system responses that the study team is examining at the time when each participant enrolls.

OTHER OUTCOMES:
Magnitude of YFV-specific Antibody Secreting Cells | Day 0 (day of vaccination), Day 3, Day 7, Day 14, Day 21, Day 28, Day 90, Day 180, Day 360
  The characterization of Yellow Fever Vaccine specific adaptive immune response will be examined as the magnitude of YFV-specific antibody secreting cells. The schedule of follow up visits depends on if participants test positive for HLA-A202 and the different immune system responses that the study team is examining at the time when each participant enrolls.
Quality of YFV-specific Antibody Secreting Cells | Day 0 (day of vaccination), Day 3, Day 7, Day 14, Day 21, Day 28, Day 90, Day 180, Day 360
  The characterization of Yellow Fever Vaccine specific adaptive immune response will be examined as the quality of YFV-specific antibody secreting cells. The schedule of follow up visits depends on if participants test positive for HLA-A202 and the different immune system responses that the study team is examining at the time when each participant enrolls.
Magnitude of YFV-specific Memory B Cells | Day 0 (day of vaccination), Day 3, Day 7, Day 14, Day 21, Day 28, Day 90, Day 180, Day 360
  The characterization of yellow fever vaccine (YFV-17D) specific adaptive immune response will be examined as the magnitude of YFV-specific memory B cells. The schedule of follow up visits depends on if participants test positive for HLA-A202 and the different immune system responses that the study team is examining at the time when each participant enrolls.
Innate immune response, Cytokines, Chemokines, Dendritic Cells, and Microarray | Day 0 (day of vaccination), Day 3, Day 7, Day 14, Day 21, Day 28, Day 90, Day 180, Day 360
  To determine the signatures of innate immune responses, cytokines, chemokines, dendritic cells, and microarray analyses for gene expression on peripheral blood mononuclear cells (PBMCs) will be examined. The schedule of follow up visits depends on if participants test positive for HLA-A202 and the different immune system responses that the study team is examining at the time when each participant enrolls.
Characterization of Epstein-Barr Virus (EBV) | Day 0 (day of vaccination), Day 3, Day 7, Day 14, Day 21, Day 28, Day 90, Day 180, Day 360
  Characterization of EBV cluster of differentiation 8 (CD8) T cells will be performed. The schedule of follow up visits depends on if participants test positive for HLA-A202 and the different immune system responses that the study team is examining at the time when each participant enrolls.
Phenotypic Analysis of Epstein-Barr Virus (EBV) | Day 0 (day of vaccination), Day 3, Day 7, Day 14, Day 21, Day 28, Day 90, Day 180, Day 360
  Phenotypic analysis of EBV CD8 T cells will be performed. The schedule of follow up visits depends on if participants test positive for HLA-A202 and the different immune system responses that the study team is examining at the time when each participant enrolls.

CONTACTS AND LOCATIONS:
Overall Officials: Rafi Ahmed, PhD, Study Chair — Emory University; Sri Edupuganti, MD, MPH, Principal Investigator — Emory University
Locations (1):
- The Hope Clinic of the Emory Vaccine Center, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Akondy RS, Monson ND, Miller JD, Edupuganti S, Teuwen D, Wu H, Quyyumi F, Garg S, Altman JD, Del Rio C, Keyserling HL, Ploss A, Rice CM, Orenstein WA, Mulligan MJ, Ahmed R. The yellow fever virus vaccine induces a broad and polyfunctional human memory CD8+ T cell response. J Immunol. 2009 Dec 15;183(12):7919-30. doi: 10.4049/jimmunol.0803903. PMID 19933869
- See also: Website for the Hope Clinic of Emory Vaccine Center — https://hopeclinic.emory.edu/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT00694655/Prot_SAP_001.pdf
  • Informed Consent Form (2024-05-31): https://cdn.clinicaltrials.gov/large-docs/55/NCT00694655/ICF_000.pdf